CLINICAL TRIAL: NCT04131699
Title: Electrical Velocimetry (ICON Cardiometry) Assessment of Hemodynamic Changes With Different Inflation Pressures During Pediatric Thoracoscopic Surgery: A Pilot Study
Brief Title: Electrical Velocimetry (ICON Cardiometry ) Assessment of Hemodynamic Changes During Pediatric Thoracoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Mohamed Abd el moneim Soaida, MD, Assistant professor, Cairo University
Other Study IDs: SMS2019-1
Record Dates: First submitted 2019-10-14; First posted 2019-10-18 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Hemodynamics
Keywords: pediatric; thoracoscopic; cardiometry; cardiac output; hemodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- pediatric thoracoscopic group: record hemodynamic changes and cardiac output at different intrathoracic pressures ( insufflation pressures 4, 5, 6 mmHg)
  Interventions: Device: Cardiotronic ICON continuous non-invasive cardiac output monitor.

INTERVENTIONS:
Device: Cardiotronic ICON continuous non-invasive cardiac output monitor. — cardiac index, cardiac output & stroke volume measured and recorded with every change in intrathoracic pressure.

SUMMARY:
Advances in endoscopic equipment and technique have led to the use of minimally invasive thoracic surgery in an increasing number of pediatric surgical procedures. Logically, thoracoscopic surgery and anesthesia can induce significant physiologic changes,, derangements of normal respiratory physiology induced by the surgical approach and the installation of carbon dioxide into the thoracic cavity can lead to alterations of normal acid-base status. Finally, surgical procedures in the chest, surgical traction or insufflation pressures impairs venous return and/or cardiac function, especially in neonates and infants. In this study Electrical Cardiometry TM (ICON, Cardiotronic/Osypka Medical, Inc., La Jolla CA, USA) is used assess the effect of different intra-thoracic pressure (insufflation pressures 4,5 & 6 mmHg) during thoracoscopic surgeries in neonates and infants on hemodynamics using electrical velocimetry (ICON) as non-invasive monitoring technique.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I-II.
2. Age neonates and infants
3. Children undergoing thoracoscopic surgery surgeries.

Exclusion Criteria:

1. Parents' or guardians' refusal.
2. Left lateral positioning
3. Congenital heart diseases.

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants and neonates who are a candidate for thoracoscopic surgeries, and suffer no congenital heart disease.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-05 (Actual)

PRIMARY OUTCOMES:
change in Cardiac index | measured before inflation, 1 minute after inflation of the thoracic cavity at 4 mm Hg, 5 mm Hg and 6 mm Hg and after deflation
  L/min/m2

SECONDARY OUTCOMES:
non invasive blood pressure | from time of induction of anesthesia and every 5 minutes and after every change in intrathoracic pressure and after deflation till end of surgery
  mmHg
heart rate | from time of induction of anesthesia and every 5 minutes and after every change in intrathoracic pressure till end of surgery
  beats per minute
stroke volume | from time of induction of anesthesia and every 5 minutes and after every change in intrathoracic pressure till end of surgery
  millilitres
systemic vascular resistance | from time of induction of anesthesia and every 5 minutes and after every change in intrathoracic pressure till end of surgery
  dynes/seconds/cm-5
cardiac output | from time of induction of anesthesia and every 5 minutes and after every change in intrathoracic pressure till end of surgery
  l/min

CONTACTS AND LOCATIONS:
Overall Officials: Sherif M Soaida, A. professor, Study Director — faculty of medicine, Cairo university, Egypt; Sara Abd EL Salam, lecturer, Study Director — faculty of medicine, Cairo university, Egypt; Maha G Hanna, professor, Study Chair — faculty of medicine, Cairo university, Egypt
Locations (1):
- Faculty of medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided